CLINICAL TRIAL: NCT02957513
Title: Improving Self-Care Decisions of Medically Underserved African-Americans With Uncontrolled Diabetes: Effectiveness of Patient-Driven Text Messaging Versus Health Coaching
Brief Title: The Management of Diabetes in Everyday Life Program
Acronym: MODEL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Tennessee (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-04735-FB; SC15-1503-28336 (Other Grant/Funding Number: PCORI)
Record Dates: First submitted 2016-10-24; First posted 2016-11-07 (Estimated); Last update posted 2019-10-10 (Actual); Status verified 2019-07

CONDITIONS: Diabetes Mellitus; Chronic Disease
Keywords: Diabetes; Uncontrolled; Chronic Disease; Chronic Conditions; Medically Underserved Areas; African Americans; Health Coaching; Health Education; Text Messaging; Text Messages; Mobile Health
MeSH Terms: conditions — Diabetes Mellitus; Chronic Disease; Health Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Text Messaging (TM) (Experimental): The TM intervention will use an extensive text message library focused on 3 key behavioral areas (diet, exercise, and medication adherence). The TM intervention will incorporate supportive cognitive behavioral strategies such as goal setting, positive reinforcement, self-talk and dealing with barriers to change. Messages will encourage social interaction (social support, problem-solving, and feedback), self-monitoring of diet and exercise, diet modification, physical activity advice and prompting and basic self- regulatory skills. Messages will be tailored based on participant demographics, health literacy, and preferences.
  Interventions: Behavioral: Text Messaging (TM)
- Health Coaching (HC) (Experimental): The HC intervention will place emphasis on the coach establishing rapport with the participant and assessing and establishing their initial goals using motivational interviewing, HC program goals, plans for future individual sessions. A written copy of personal health goals will be given to patients at the end of the first session. Coaches will aim to meet with participants for individual HC sessions bi-monthly the first 2-3 months followed by monthly for 8 - 9 months to provide information and support regarding health habits focusing sessions on areas related to patient-identified health goals, needs, and barriers to change. Sessions can occur in person or by phone based on patient preference.
  Interventions: Behavioral: Health Coaching (HC)
- Enhanced Usual Care (EC) (Active Comparator): All participants in all 3 study arms (TM, HC, and EC) will receive enhanced usual care. Usual care in the participating practices will be supplemented through the following key EC resources:
  A. Patient-focused Resources including: 1) MODEL Program Toolkit, and 2) low literacy diabetes educational materials.
  B. Availability of diabetes support services including: 1) peer group support sessions, 2) diabetes education, 3) MyDiabetesCenter.org resources, and 4) Diabetes Coalition education hub resources.
  C. Practice-focused components including: 1) practice training/continuing medical education, and 2) reporting of diabetes performance measures.
  Interventions: Behavioral: Text Messaging (TM); Behavioral: Health Coaching (HC); Behavioral: Enhanced Usual Care (EC)

INTERVENTIONS:
Behavioral: Text Messaging (TM) — As specified in the arm description above
  Arms: Enhanced Usual Care (EC); Text Messaging (TM)
Behavioral: Health Coaching (HC) — As specified in the arm description above
  Arms: Enhanced Usual Care (EC); Health Coaching (HC)
Behavioral: Enhanced Usual Care (EC) — As specified in the arm description above
  Arms: Enhanced Usual Care (EC)

SUMMARY:
The overall goal of this study is to compare how well motivational messages (text messages from the doctor's office), diabetes health coaches, and enhanced usual care with diabetes education materials (provided at the doctor's office) work to help African-American adults with uncontrolled diabetes improve their diabetes self-care decisions. Self-care is difficult when you have diabetes, especially when patients have other medical conditions, their diabetes is uncontrolled, and when they live in an area without many primary care doctors. Many studies have show that encouraging text messages from the doctor's office and health coaches can help people take better care of themselves. But before primary care clinics around the country start trying to send texts, hire health coaches, or provide additional educational materials it is critical for them to know which approach is more likely to help.

This study will assign African-American diabetics to either text messages, health coaches, or enhanced care to find out which one works better. The investigators especially want to find out if one works better for people at highest risk. Lastly, the investigators want to find out if messages or coaches help people improve their blood sugar, quality of life, and their feelings about primary care.

The study will test messages, coaches, and enhanced care side by side in primary care doctors' offices. The messaging and coaching programs will give patients pretty much the same information, but in different ways. The text messages will be written carefully based on each patient's needs and interests. The coaches will be trained in how to help people get motivated and work to reach their health goals.

This study will include 646 African-American adults, ages 18 and above, with uncontrolled diabetes and one or more additional chronic condition, living in medically underserved communities. People will have to have a cell phone or smart phone with texting capability and be able to use it to participate. 258 participants will get messages, 258 will get coaches, and 130 will receive enhanced care.

The investigators will be able to tell if messages and coaches work by seeing if people improve their diabetes self-care decisions, and if their blood sugar, quality of life, and feelings about primary care get better. The long-term study goal is to get primary care clinics all over the country to start using motivational messages or health coaches if they work well.

DETAILED DESCRIPTION:
Background and Significance: There is a critical need to determine the comparative effectiveness of text messaging (TM) and health coaching (HC) among African-Americans with uncontrolled diabetes and multiple chronic conditions living in medically underserved areas (MUA) and to identify which modality yields greater improvement in diabetes self-care at-risk urban and rural subpopulations. Although numerous recent studies demonstrate the effectiveness of either TM or HC in improving diabetes and other chronic disease self-care behaviors, and to the knowledge of the investigators no information is available regarding comparative effectiveness of these modalities in urban and rural subgroups. Prevalence of diabetes, related comorbidities, poverty, obesity, food insecurity, and tobacco use is higher in rural areas as compared with urban. Moreover, rural areas struggle to address these needs because of lower access to transportation, primary care, specialty care, diabetes education, and mental health resources. However, urban living has its own unique set of problems-including increased stress and fear for one's physical safety-that may impact the comparative effectiveness of HC and TM. Although there are HC studies that show effectiveness in interventions either in rural or urban areas, there are no HC studies of which the investigators are aware that specifically examine the differences in U.S. rural and urban participants in regards to engagement rates and clinical outcomes from a health coaching intervention. Similarly, telemedicine and mobile health approaches have been particularly advocated for rural populations yet little evidence supports their comparative benefit. The lack of comparative effectiveness of text messaging and health coaching for diabetes self-care in vulnerable urban and rural subgroups represents a critical gap in research that the study is designed to directly address. The study will compare both strategies with enhanced usual care (EC) with diabetes educational materials.

Study Aims: As a result, this research will use a pragmatic randomized trial to determine the comparative effectiveness of patient-driven TM versus HC versus EC for African-American adults with uncontrolled diabetes and multiple chronic conditions in MUA with an emphasis on identifying and quantifying important interactions between key baseline characteristics and treatment arm. Specific aims include: Aim 1-Quantify the effectiveness of TM, HC, and EC in improving the primary outcome measures (diabetes self-care activities related to general diet, exercise and medication adherence); Aim 2-Determine the contributions of six key, baseline patient characteristics: 1) urban vs. rural residence, 2) health literacy, 3) medical complexity, 4) social complexity, 5) smart vs. cell phone ownership, and 6) age, to the comparative effectiveness of TM, HC, and EC; and Aim 3-Quantify the effectiveness of TM, HC, and EC in improving secondary outcomes of average blood sugar, quality of life, and primary care engagement. The long-term objectives are to disseminate and foster implementation of the results of this research in MUA nationwide to improve critical self-care supports in primary care for our most vulnerable populations.

Overall study design: Pragmatic randomized clinical trial.

Main components of the intervention and comparator(s): The study will test two critical strategies for patient engagement that may lead to substantive improvements in the quality of care and outcomes most important to vulnerable patients with diabetes: 1) patient-driven TM, and 2) patient-driven HC. The two parallel primary care-based and patient-driven study interventions (i.e. TM and HC) have been designed to provide approximately the same content, but with two alternative delivery mechanisms. TM will incorporate supportive cognitive behavioral strategies to encourage improved diabetes self-care decisions and will be tailored based on participant demographics, health literacy, preferences, treatment self-regulation, perceived competency and reported barriers to self-care. Motivational interviewing focused HC will aim to meet with participants for individual HC sessions bi-monthly the first 2 months (Intensive Phase-4 sessions following randomization) followed by monthly for remaining 8 months (12 sessions total) to provide support regarding diet/weight loss, physical activity, and medication adherence tailored according to patient-identified health goals. Both strategies will be compared with EC with diabetes educational materials.

Study population: For the main comparative effectiveness analysis (Aim 1) the total sample size (after dropouts) is N=800 with 40% randomized to the TM arm (N1=320), 40% to the HC arm (N2=320), and 20% to the EC arm (N3 = 160). Participants include African-American adults, ages 35-75, with uncontrolled diabetes and multiple chronic conditions, living in medically underserved communities in the MidSouth who have a cell phone or smart phone with texting capability and complete a two-week run-in period demonstrating responsiveness to TM.

Primary/secondary outcomes: The primary outcome measures assessing effectiveness include: three (out of six total) subscales of the revised Summary of Diabetes Self-Care Activities questionnaire assessing general diet, exercise, and medication adherence. Secondary outcomes include: diabetes-specific quality of life using the Diabetes-39, primary care engagement using National Health Interview Survey questions regarding delayed needed care, and average blood sugar (A1c) obtained from medical records and reported in the DWPC-R.

Analytic methods: For Aim 1, in the context of repeated measures ANOVA, using t-tests within arm to detect change from baseline to 12-months (Follow-up 3), power exceeds 0.9 for all primary outcomes. For Aim 2, six analyses will assess heterogeneity of treatment effects by evaluating the interaction of each key, dichotomized, baseline characteristic with treatment arm, estimating means and standard errors of six subclasses, and within each characteristic (e.g. low or high health literacy) testing for differences between TM and HC, TM and EC, and HC and TM. Analyses for Aim 3 will be conducted as described above for Aim 1.

ELIGIBILITY:
Inclusion Criteria:

* self-identified African-American adults
* diagnosis of uncontrolled diabetes (HbA1C > 8)
* have at least one other of 13 chronic health conditions (hypertension, congestive heart failure, coronary artery disease, cardiac arrhythmias, hyperlipidemia, stroke, arthritis, asthma, cancer, chronic kidney disease, chronic obstructive pulmonary disease, depression, and osteoporosis and excluding dementia)) using the CMS ICD-9-CM-based definitions
* is receiving or will receive care at one of our identified clinical sites
* has a cell phone or smart phone with texting and voicemail capabilities
* is not planning to move from the area in the next year
* is able to provide informed consent
* is English speaking
* completes a two-week run-in period for text message and voice message use

Exclusion Criteria:

* inability to understand consent procedures
* Pregnant
* presence of an unstable psychiatric condition or dementia
* perceived unwillingness or inability to participate
* inability to successfully complete the text message and voice message screening test
* Plans to move from the area and change primary care physicians in the next year.
* Diagnosis of severe depression in the last six months
* Individuals with cognitive impairment will be excluded if they experience difficulty either understanding, following directions, or communicating clearly with program staff. Individuals will be excluded if they exhibit uncontrolled psychiatric symptoms and/or behaviors that may present a danger to program staff or to the study participants themselves.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 646 (Estimated)
Dates: Start 2016-11-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Diabetes Self-Care Activities | 1 year
  The Revised Summary of Diabetes Self-Care Activities Questionnaire (SDSCA) assesses DM self-care over the previous 7 days for 7 core behaviors: smoking, diet, exercise, blood sugar testing, foot care, smoking, and medication adherence (12 items)

SECONDARY OUTCOMES:
Diabetes-Specific Quality of Life | 1 year
  The Diabetes-39 has 5 domains: DM control, Anxiety and worry, Social burden, Sexual functioning, and Energy and mobility
Primary Care Engagement | 1 year
  Selected National Health Interview Survey (NHIS) questions assess 3 primary domains: (a) Usual source of care when sick; (b) Usual source of preventive care; and (c) Delay in needed care
Quality of Care | 1 year
  The Patient Assessment of Chronic Illness Care (PACIC) measures specific actions or qualities of care based on Chronic Care Model
Average Blood Sugar (A1c) | 1 year
  The Hemoglobin A1c blood test assesses average blood sugar over the past 6 weeks to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: James E Bailey, MD, MPH, Principal Investigator — University of Tennessee
Locations (19):
- United States (19):
  - Hawkins Family Medicine, Holly Springs, Mississippi
  - Covington Pike Primary Care, Methodist Le Bonheur Healthcare, Bartlett, Tennessee
  - Tipton Family Medicine Center, Covington, Tennessee
  - University of Tennessee Family Practice Center, Jackson, Tennessee
  - Eastmoreland Internal Medicine, Memphis, Tennessee
  - Midtown Internal Medicine, Methodist Le Bonheur Healthcare, Memphis, Tennessee
  - Peabody Family Care, Methodist Le Bonheur Healthcare, Memphis, Tennessee
  - UT Methodist Physicians, Eastmoreland Endocrinology, Memphis, Tennessee
  - Christ Community Health Services - Third Street Health Center, Memphis, Tennessee
  - TriState Medical Group PLLC, Memphis, Tennessee
  - Motley Internal Medicine, Methodist Le Bonheur Healthcare, Memphis, Tennessee
  - South Internal Medicine, Methodist Le Bonheur Healthcare, Memphis, Tennessee
  - UT Methodist Physicians, South Endocrinology, Memphis, Tennessee
  - PennMarc Internal Medicine, Methodist Le Bonheur Healthcare, Memphis, Tennessee
  - Christ Community Health Services, Broad Avenue Health Center, Memphis, Tennessee
  - Memphis Health Center, Memphis, Tennessee
  - Christ Community Health Center - Raleigh Health Center, Memphis, Tennessee
  - Whitney Slade Internal Medicine, Methodist Le Bonheur Healthcare, Memphis, Tennessee
  - Regional One Health, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Data may be exported from the database system that houses study data in a variety of formats for sharing and/or analysis. At study completion, the investigators anticipate extracting all data from the system for sharing with other sources once appropriate governance and sharing restrictions have been addressed. Data dictionaries and associated metadata will be provided as needed upon request. Data can be shipped or mailed in approved, encrypted format or collected via SFTP (secure file transfer protocol) from our servers. The cost of allowing prospective investigators access to the de-identified data from this project will include IRB costs to review the application, salary support to cover staff time to review the concept proposal, submit documents to the IRB, and to establish password-protected and secured transfer application of the data. This cost is per application per investigator who wishes access granted to the de-identified data.

REFERENCES:
- [Derived] Bailey JE, Surbhi S, Gatwood J, Butterworth SW, Coday M, Chen M, Gutierrez ML, Shuvo SA, Brooks IM, Binkley BL, Riordan CJ, Steinberg HO, Leak CL, Breen WR Jr, Dowell SW, Tolley EA. Comparative Effectiveness of Diabetes Self-Care Interventions in African-American Adults: A Three-Arm Randomized Controlled Trial. J Gen Intern Med. 2025 Oct 20. doi: 10.1007/s11606-025-09882-z. Online ahead of print. PMID 41116096
- [Derived] Tolley EA, Surbhi S, Bailey JE. Using preliminary data and prospective power analyses for mid-stream revision of projected group and subgroup sizes in pragmatic patient-centered outcomes research. Data Brief. 2020 Nov 17;33:106529. doi: 10.1016/j.dib.2020.106529. eCollection 2020 Dec. PMID 33304950
- [Derived] Bailey JE, Surbhi S, Gatwood J, Butterworth S, Coday M, Shuvo SA, Dashputre AA, Brooks IM, Binkley BL, Riordan CJ, Steinberg HO, Gutierrez ML, Haley LE, Leak CL, Tolley EA. The management of diabetes in everyday life study: Design and methods for a pragmatic randomized controlled trial comparing the effectiveness of text messaging versus health coaching. Contemp Clin Trials. 2020 Sep;96:106080. doi: 10.1016/j.cct.2020.106080. Epub 2020 Jul 9. PMID 32653539
- [Derived] Gatwood J, Shuvo S, Ross A, Riordan C, Smith P, Gutierrez ML, Coday M, Bailey J. The Management of Diabetes in Everyday Life (MODEL) program: development of a tailored text message intervention to improve diabetes self-care activities among underserved African-American adults. Transl Behav Med. 2020 Feb 3;10(1):204-212. doi: 10.1093/tbm/ibz024. PMID 30794316
- See also: PCORI Project Summary — http://www.pcori.org/research-results/2016/improving-self-care-decisions-medically-underserved-african-americans